CLINICAL TRIAL: NCT07137819
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Adaptive Phase 3 Study to Evaluate the Efficacy and Safety of Sinecatechins (Defined Extract of Green Tea Leaves) Ointment in Adult Patients With Actinic Keratosis of the Scalp and the Face
Brief Title: Phase 3 - Evaluation of Veregen® 10% Ointment as New Herbal Topical Treatment for Actinic Keratosis
Acronym: EXACT-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aresus Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-502811-12-00 - Pro_VER-01; 2022-502811-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Actinic Keratosis of Face and Scalp
Keywords: Veregen® 10% ointment; Actinic Keratosis (AK) of the Scalp and/or the Face; Germany; Sinecatechins; Green tea
MeSH Terms: conditions — Keratosis, Actinic | interventions — Therapeutics; green tea extract polyphenone E; Ointments

STUDY DESIGN:
Intervention Model Description: The primary objective of the study is to show superiority of Veregen® 10% ointment to Placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum arm using Veregen® 10% ointment (Experimental): This arm uses Veregen® 10% ointment to measure complete (100%) clearance of a pre-defined treatment area (TA) following a treatment period of 12 weeks and a 4-weeks post-treatment (PT) period (i.e., after 16 weeks at most in patients without complete clearance at the end of the treatment (EoT) period).
  Interventions: Drug: Topical treatment
- Placebo arm using placebo to Veregen® 10% ointment (Placebo Comparator): This arm uses placebo ointment for self-treatment of patients in a pre-defined treatment area (TA) following a treatment period of 12 weeks and a 4-weeks post-treatment (PT) period (i.e., after 16 weeks at most in patients without complete clearance at the end of the treatment (EoT) period).
  Interventions: Drug: Topical treatment

INTERVENTIONS:
Drug: Topical treatment — Self-treatment of patients with ointment of a pre-defined treatment area (TA) following a treatment period of 12 weeks and a 4-weeks post-treatment (PT) period (i.e., after 16 weeks at most in patients without complete clearance at the end of the treatment (EoT) period).
  Other Names: Veregen 10% ointment

SUMMARY:
The goal of this clinical trial is to show superiority of Veregen® 10% ointment to Placebo measured by complete (100%) clearance of a pre-defined treatment area (TA) following a treatment period of 12 weeks and a 4-weeks post-treatment (PT) period (i.e., after 16 weeks at most in patients without complete clearance at the end of the treatment (EoT) period).

DETAILED DESCRIPTION:
Participants type: Patients Age range: 18-64 years, 65+ years; male and female Locations: Germany

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate, obtained written informed consent.
* Male or female patients ≥ 18 years.
* Clinically confirmed diagnosis of mild to moderate Actinic keratosis (AK) of the face including the forehead (excluding eyelids, lips and mucosa) and/or the bald scalp.
* Presence of at least 4 but not more than 8 isolated (i.e. discrete and quantifiable) AK lesions located in a contiguous treatment area (TA) on the face and/or bald scalp of 25 square-cm.
* AK lesions of the TA must be clinically typical AK lesions of Olsen grade I and/or grade Olsen grade II.
* Ability to follow study instructions and likely to complete all study requirements.

Exclusion Criteria:

* TA is within 5 cm of an incompletely healed wound or infected area of the skin.
* Patients not willing to abstain from sunbathing (including solarium) or any outdoor activities with intensive sun exposure without taking appropriate measures to protect the treatment areas during the study.
* Patients with a tendency to manipulate skin parts e.g. scratching.
* Pregnant or breast-feeding patients.
* Patients currently or within the past 4 weeks participating in another clinical study.
* Any previous randomization into this clinical study.
* Any suspicion of current drug and/or alcohol abuse.
* Patient is institutionalized because of legal or regulatory order.
* Dependency (as an employee or relative) to the sponsor/responsible CRO or investigator.
* Any condition that in the opinion of the investigator can influence the evaluation of the treatment, and other assessments.
* Hypersensitivity, intolerance or allergies against ingredients of Veregen® 10% ointment and/or Placebo ointment.
* AK lesions in the TA with atypical clinical appearance (e.g. TA contains massively hyperkeratotic and hypertrohic lesions (Olsen grade III AK), recalcitrant lesions, cutaneous horns, and/or lesions that had not responded to 2 previous cryotherapies).
* Have received the following topical or physical treatments for any indication in the treatment area within the designated time period before treatment with study drug: a) Curettage, Photodynamic therapy, Topical inhibitors of Src tyrosine kinase signaling and tubulin polymerization (e.g.,Tirbanibulin) for/in a period of 12 weeks; b) Topical retinoids, Topical diclofenac preparations, Topical 5-fluorouracil preparations, Topical immunomodulators (e.g., Imiquimod) for/in a period of 6 weeks; c) Topical steroids, Cryo-, thermo- or chemodestruction, Surgical excision for/in a period of 4 weeks.
* Initiation of treatment with the following systemic treatments for any indication within 2 weeks before Baseline: Immunomodulators or immunosuppressive therapies, Diclofenac, Corticosteroids (oral or injectable), Inhaled corticosteroids (>1200 µg/day for beclomethasone, or >600 µg/day for fluticasone)
* Current or planned intake of high dosed oral green tea preparations for any reason
* Current or planned application of dermal preparations with astringent effect on the TA, such as zinc paste or tannin-containing ointments/creams
* Patients taking a drug with known potential for skin reactions must have taken it at a stable dose for at least 2 weeks prior to Baseline, except in cases where no previous skin reactions have occurred at any dose.
* Women of childbearing potential (WOCBP) will not be considered unless they use a highly effective method of contraception (failure rate of less than 1% per year) during the interventional period until 4-weeks PT (EoI, V9).
* Within the TA, any suspicion of other malignant or benign skin tumors.
* History of a genetic skin-cancer disorder (e.g. xeroderma pigmentosum) and/or invasive tumor in the TA, such as a Merkel cell tumor, an invasive spinocellular carcinoma or a BCC (Basal Cell Carcinoma) and/or any skin cancer (suspected or diagnosed recently or within 5 years ago before screening).
* History or evidence of skin conditions other than AK that would interfere with evaluation of the study medication (e.g. eczema, unstable psoriasis).
* Patients having any significant physical abnormalities in the TA that may cause difficulty with examination or AK assessments (e.g. tattoes, scars, hyperpigmentation, etc.).
* Evidence of clinically significant or unstable medical conditions such as: (a) metastatic tumor or tumor with high probability of metastatic spread, (b) heart failure (NYHA class III or higher), (c) immunosuppressive disorder (e.g. HIV, organ transplant patients), (d) hematologic, hepatic, renal, neurologic or endocrine disorder, (e) collagen-vascular disorder (e.g. cerebro-vascular or other bleeding disorder), (f) gastrointestinal disorder (e.g. active ulcera or history of recurrent peptic ulcera or hemorrhage).
* Patients not willing to stop using skin care products (e.g. self-tanning products, sunscreens, make-ups/colored day care cremes, topical treatments with anti-aging products, vitamin A, vitamin C, and/or vitamin E containing ointments and gels) in the TA during the interventional period of the study (i.e., during the treatment and until 4 weeks post-treatment).
* Patients not willing to stop any use of make-ups colored day care cremes, and sunscreens in the treatment area within 12 hours prior to an on-site visit during the PTFU period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Primary objective is to show superiority of Veregen® 10% ointment to Placebo measured by complete (100%) clearance of a pre-defined treatment area (TA) following a treatment period of 12 weeks and a 4-weeks post-treatment (PT) period. | From enrollment to the end of treatment period at 12 weeks and a 4-weeks post-treatment (PT) period (i.e., after 16 weeks).
  The primary objective of the study is to show superiority of Veregen® 10% ointment to Placebo measured by complete (100%) clearance of a pre-defined treatment area (TA) following a treatment period of 12 weeks and a 4-weeks post-treatment (PT) period (i.e., after 16 weeks at most in patients without complete clearance at the end of the treatment (EoT) period).

CONTACTS AND LOCATIONS:
Locations (1):
- Aresus Pharma GmbH, Strausberg, Germany